CLINICAL TRIAL: NCT02379429
Title: Care of the Urothelial Cancer Patient and Prospective Collection of Biospecimens From Healthy Volunteers and Urothelial Cancer Patients
Brief Title: Care of the Urothelial Cancer Patient and Prospective Procurement of Urothelial Cancer Tissue
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150087; 15-C-0087
Record Dates: First submitted 2015-03-04; First posted 2015-03-05 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11-13

CONDITIONS: Bladder Cancer; Urinary Tract Cancer; Urothelial Cancer; Healthy Volunteers
Keywords: Specimen Collection; Urine; Blood; Saliva; Natural History
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Participants: Adults with biopsy-proven or suspected urothelial cancer who require diagnostic or therapeutic intervention
- 2/Healthy Volunteers: Healthy volunteers from whom blood, saliva and urine samples are easily obtainable.

SUMMARY:
Background:

Urothelial cancer is cancer of the bladder, ureter, and urethra. Researchers want to better understand what changes in a person s cells and genes cause this cancer to form. This may help them find new ways to treat it.

Objective:

- To perform DNA sequencing to help researchers learn the differences between normal tissue and tumor tissue. Also, to learn how molecular changes - including gene changes - might help predict the course of disease and how people respond to therapy.

Eligibility:

- Adults age 18 and older who have or are suspected of having urothelial cancer or an inherited disorder that raises their risk of getting bladder cancer.

Design:

* Participants will be screened with a physical exam. Their medical records and tissue samples will be reviewed.
* Eligible participants will give tissue blocks of their original tumor. The blocks will be put in a tissue bank.
* Participants medical records may be reviewed.
* Participants may have a medical history and physical exam.
* Participants may have blood and urine tests. They may have imaging scans. They may give urine, blood, and saliva samples. These samples may be used in future research.
* If participants need surgery for their cancer, researchers will keep some of the tissue (both tumor and normal tissue). The tissue may be used in future research.
* Participants will go back to the Clinical Center in 6 months. They may give saliva, urine, and blood samples. After 6 months, they will be seen by their local doctor for standard post-surgical visits.
* Participants will be called every 6 months to give health updates.

DETAILED DESCRIPTION:
Background:

* Urothelial carcinoma, present as lower or upper urinary tract disease, is the most expensive malignancy to treat from diagnosis to death, and no major advances in drug therapy have taken place in the last two decades.
* Understanding the molecular mechanisms and genomic alterations that cause urothelial carcinoma will provide the foundation for the development of novel targeted therapeutic agents for this disease. Since 1982 investigators in the Urologic Oncology Branch have been studying the genetic basis of urologic cancers. The identification of the genes for cancer of the kidney has led to the approval by the FDA of a number of new agents for patients with advanced disease. Similarly, it is our goal to study the cancer biology (genomic, molecular, and cellular biology) of urothelial carcinoma in order to develop novel treatment strategies.
* Collection of patient tumor samples allows us to study molecular and biologic pathways and develop novel targeted therapies. Correlation of these samples with clinical outcomes in patients allows us to predict and understand clinical outcomes and possibly develop predictive and/or prognostic biomarkers.
* Collection of blood, urine and saliva from healthy volunteers will allow us to distinguish normal and inflammatory conditions from malignant diseases. Furthermore, the specimens will provide appropriate controls for comparison.

Objective (Primary):

* Collect blood, urine, and benign and malignant tissue from patients with known or suspected urothelial cancer for the purpose of elucidating the molecular mechanisms of carcinogenesis in urothelial cancer and ultimately, identifying novel therapeutic targets.
* Collect blood, urine and saliva from healthy volunteers for the purpose of establishing controls for comparison with urothelial cancer specimens.

Eligibility:

* Adults with biopsy-proven or suspected urothelial cancer who require diagnostic or therapeutic intervention as part of their diagnosis, standard of care treatment, or followup/surveillance for their neoplasm.
* Healthy volunteers from whom blood, saliva and urine samples are easily obtainable.

Design:

* Care of the patient with urothelial carcinoma will be provided as per medically indicated standards and in the process, normal and malignant urothelial cancer tissues may be obtained at the time of clinically indicated diagnostic and/or therapeutic intervention.
* Blood, urine, and saliva samples for research may be obtained from patients and healthy volunteers at baseline. Additionally, blood and urine may be collected from patients at follow-up intervals.
* No investigational or experimental therapy will be given as part of this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA FOR UROTHELIAL CANCER PARTICIPANTS:
* Adults (>= 18 years of age) with biopsy-proven or suspected urothelial cancer who require and are willing to undergo diagnostic or therapeutic intervention as part of their diagnosis, standard of care treatment, or follow-up/surveillance for their neoplasm.
* ECOG performance status of 0-3.
* Must be willing and able to provide informed consent.

EXCLUSION CRITERIA:

* Subjects who are pregnant.
* Subjects co-morbidities preclude diagnostic or therapeutic intervention. Co-morbidities include:

  --Ongoing treatment for another non-skin malignancy.
* History of hepatitis B/C or HIV. Patients who are HIV positive are excluded from this study because treatment with immunomodulatory agents for immunosuppressed patients would affect sample analysis and skew the data.

ELIGIBILITY CRITERIA FOR HEALTHY VOLUNTEERS

INCLUSION CRITERIA:

-Adults (greater than or equal to 18 years of age) and able to give informed consent.

EXCLUSION CRITERIA:

* Subjects who are pregnant.
* Diagnosis of cancer requiring treatment other than minor resection of basal cell or squamous cell skin cancers.
* Heart, lung, kidney disease, or other medical conditions as per Principal Investigator discretion.
* History of acute or chronic hepatitis B/C or HIV infection. Patients who are HIV positive are excluded from this study because treatment with immunomodulatory agents for immunosuppressed patients would affect sample analysis and skew the data.
* Healthy volunteers who are family members with germline mutations.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two different groups of population: 1. Adults age 18 and older who have or are suspected of having urothelial cancer or an inherited disorder that raises their risk of getting bladder cancer 2. Healthy volunteers (18 and older),the specimens will provide appropriate controls for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-11-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Collect samples for the purpose of studying the molecular mechanisms of carcinogenesis in urothelial cancer. | ongoing
  Collection of blood, urine, saliva, and/or benign and malignant tissue

SECONDARY OUTCOMES:
Perform molecular profiling and analysis to better characterize urothelial cancer and identify novel targets. | ongoing
  Collection of blood, urine, saliva, and/or benign and malignant tissue
Develop stable urothelial / bladder cancer cell lines from procured tissue when feasible. | ongoing
  Generating cell lines
Collect detailed history, pathologic data, perioperative findings, and treatment data to better characterize the natural and clinical histories of urothelial cancer when feasible. | ongoing
  Collection of clinical histories of urothelial cancer

CONTACTS AND LOCATIONS:
Overall Officials: Raju R Chelluri, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-C-0087.html